CLINICAL TRIAL: NCT05561751
Title: A Phase 2, Randomized, Open-Label Study to Assess the Safety and Efficacy of GPC 100 and Propranolol With and Without G-CSF for the Mobilization of Stem Cells in Patients With Multiple Myeloma Undergoing Autologous Stem Cell Transplant
Brief Title: Ph2, Study to Assess the Safety and Efficacy of GPC 100 and Propranolol With and Without G-CSF for the Mobilization of Stem Cells in Patients With Multiple Myeloma Undergoing Autologous Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GPCR Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPC-100-001
Record Dates: First submitted 2022-09-26; First posted 2022-09-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Propranolol; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: This is a randomized, open-label study. Patients will be screened within 28 days prior to the study drug administration. Patients will be randomly assigned to 1 of 2 treatment arms prior to study drug administration.
  Approximately 40 patients will be randomized in a 1:1 ratio to the following treatment arms:
  * GPC-100 in combination with propranolol; or
  * GPC-100 in combination with propranolol and G-CSF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GPC-100 in combination with propranolol; (Experimental): Patients will be randomly assigned to 1 of 2 treatment arms prior to study drug administration.
  Approximately 40 patients will be randomized in a 1:1 ratio to the following treatment arm:
  • GPC-100 in combination with propranolol; or
  Interventions: Drug: GPC-100; Drug: Propranolol
- GPC-100 in combination with propranolol and G-CSF (Experimental): Patients will be randomly assigned to 1 of 2 treatment arms prior to study drug administration.
  Approximately 40 patients will be randomized in a 1:1 ratio to the following treatment arm:
  • GPC-100 in combination with propranolol and G-CSF.
  Interventions: Drug: GPC-100; Drug: Propranolol; Drug: G-CSF

INTERVENTIONS:
Drug: GPC-100 — GPC-100 is to be administered at a dose of 3.14 mg/kg GPC-100 free base via IV infusion. The corresponding volume of the reconstituted GPC-100 solution calculated based on the patient weight will be administered via IV infusion over 15 min
Drug: Propranolol — propranolol
Drug: G-CSF — G-CSF
  Arms: GPC-100 in combination with propranolol and G-CSF

SUMMARY:
This is a randomized, open-label study. Patients will be screened within 28 days prior to the study drug administration. Patients will be randomly assigned to 1 of 2 treatment arms prior to study drug administration.

Approximately 40 patients will be randomized in a 1:1 ratio to the following treatment arms:

* GPC-100 in combination with propranolol; or
* GPC-100 in combination with propranolol and G-CSF. To characterize the safety and clinical activity of GPC-100, the study will employ a Bayesian Optimal Phase II (BOP2) design to enroll patients for each arm.

All patients will receive via IV 3.14 mg/kg GPC-100 (Burixafor) at least 2 hours prior to leukapheresis sessions from Days 7-8 (Days 9-11 optional) and 30 mg propranolol (3 x 10 mg tablets) twice daily at 8:30 AM (+/- 1 hr) and 4:00 PM (+/- 1 hr) local time from Days 1 to 8 (and on Days 9-11, if applicable). Patients will administer the first dose of propranolol onsite on Day 1. Patients will be provided with doses of propranolol for self-administration at time points when they are not otherwise required to be onsite. Sites should contact patients via telephone to confirm propranolol administration for doses administered outside of clinic.

DETAILED DESCRIPTION:
This is a randomized, open-label study. Patients will be screened within 28 days prior to the study drug administration. Patients will be randomly assigned to 1 of 2 treatment arms prior to study drug administration.

Approximately 40 patients will be randomized in a 1:1 ratio to the following treatment arms:

* GPC-100 in combination with propranolol; or
* GPC-100 in combination with propranolol and G-CSF. To characterize the safety and clinical activity of GPC-100, the study will employ a Bayesian Optimal Phase II (BOP2) design to enroll patients for each arm.

All patients via IV 3.14 mg/kg GPC-100 (Burixafor) at least 2 hours prior to leukapheresis sessions from Days 7-8 (Days 9-11 optional) and 30 mg propranolol (3 x 10 mg tablets) twice daily at 8:30 AM (+/- 1 hr) and 4:00 PM (+/- 1 hr) local time from Days 1 to 8 (and on Days 9-11, if applicable). Patients will administer the first dose of propranolol onsite on Day 1. Patients will be provided with doses of propranolol for self-administration at time points when they are not otherwise required to be onsite. Sites should contact patients via telephone to confirm propranolol administration for doses administered outside of clinic.

Only patients randomized to the treatment arm receiving GPC-100 in combination with propranolol and G-CSF will receive SC injections of 10 microgram/kg/day G-CSF at 5:00 PM (+/- 3 hr) local time on Days 3 to 7. Patients in this arm will receive G-CSF injections on Days 8-10 at 5:00 PM (+/- 3 hr) local time only if they will undergo the optional third-fifth days of mobilization/collection (Days 9-11) at the Investigator's discretion.

On Days 7 and 8 (and on Days 9-11, if applicable), the patient will receive a morning 30 mg propranolol dose (3 x 10 mg tablets) followed immediately by a 3.14 mg/kg dose of GPC-100 free base (active ingredient) and will start collection of CD34+ stem cells via leukapheresis.

ELIGIBILITY:
Inclusion Criteria

To be eligible to participate in this study, patients must meet all the following criteria:

1. Male or female, greater than or equal to18 years of age;
2. Patients with diagnosis of MM per the International Myeloma Working Group criteria ;
3. Eligible for ASCT at the Investigator's discretion;
4. >4 weeks since completion of last cycle of chemotherapy prior to Day 1;
5. Patient must be on first or second complete response or partial response;
6. Eastern Cooperative Oncology Group performance status of 0 or 1 (see Appendix C);
7. Systolic blood pressure (SBP) 100 - 160 mmHg inclusive, and diastolic blood pressure (DBP) 60 - 100 mmHg inclusive;
8. ANC greater than or equal to1.0 x 109/L on Screening laboratory assessments;
9. Platelet count greater than or equal to100 x 109/L on Screening laboratory assessments;
10. Creatinine clearance greater than or equal to 30 ml/min, as calculated according to the Cockcroft-Gault formula;
11. Aspartate aminotransferase and alanine aminotransferase less than or equal to 2 x upper limit of normal (ULN) and total bilirubin less than or equal to1.5 x ULN on Screening laboratory assessments;
12. Adequate cardiac (left ventricular ejection fraction [LVEF] greater than or equal to 50%) and pulmonary function (room air O2 saturation value greater than or equal to 92%);
13. For females, 1 of the following criteria must be fulfilled:

    1. At least 1 year postmenopausal; or
    2. Surgically sterile, or willing to use a double-barrier method of contraception (e.g., intrauterine device plus condom, spermicidal gel plus condom) from Day 1 until 28 days after the last dose of GPC-100.
14. Males must be willing to use a reliable form of contraception (e.g., use of a condom or a partner fulfilling the above criteria) from Day 1 until 28 days after the last dose of GPC-100; and
15. Patients must be willing and able to provide signed informed consent. 4.2 Exclusion Criteria

Patients must be excluded if they meet any of the following criteria:

1. greater than or equal to 25% of BM irradiated within 5 years prior to Day 1 (see Appendix D);
2. No more than one year of therapy administered prior to stem cell mobilization, per institution standards;
3. Patients who have undergone previous stem cell transplant;
4. Receipt of G-CSF within 2 weeks prior to Day 1;
5. History of another malignancy except for the following:

   1. Adequately treated local basal cell or squamous cell carcinoma of the skin;
   2. Adequately treated carcinoma in situ of the cervix without evidence of disease;
   3. Adequately treated papillary, noninvasive bladder cancer; or
   4. Low-grade prostate cancer that is on active surveillance and not expected to clinically progress over 2 years.
6. Patients who are on BBs and unable to switch therapy; Note: Patients on BBs who are able to switch therapy will undergo a gradual tapering of their current BB under the guidance of the Investigator. At the Investigator's discretion, the initial days of propranolol administration may be permitted to overlap with the final days of tapering of the previous BB. Patients may not be treated with cardiovascular drugs that would interact with propranolol including angiotensin-converting enzyme (ACE) inhibitors, calcium channel blockers, and alpha blockers at study enrollment and while on propranolol during the study.
7. Patients with severe asthma who require beta agonist therapy;
8. History of poor and uncontrolled cardiovascular or pulmonary disease such as myocardial infarction, cardiac arrhythmias, transient ischemic attack, congestive heart failure (New York Heart Association heart failure class >2), stroke, unexplained syncope, or chronic obstructive pulmonary disease;
9. History of long QT syndrome or torsade de pointes;
10. Patients with a QTcF >470 msec or PR interval >280 msec on Screening 12-lead electrocardiogram (ECG);
11. Active infection requiring treatment in the 7 days before Day 1;
12. Positive polymerase chain reaction test from nasal specimen for SARS-CoV-2 within 7 days prior to Day 1;
13. Pregnant or breastfeeding;
14. Known psychiatric or substance abuse disorder that would interfere with Protocol compliance;
15. Receipt of any other investigational drug or device within 1 month before Day 1; or
16. Receipt of prior treatment with CXCR4 inhibitor for stem cell collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients that achieve >=2 x 10^6 CD34+ cells/kg in 2 leukapheresis sessions | 2 days
  Determine the proportion of patients that will achieve >=2 x 10^6 CD34+ cells/kg in 2 leukapheresis sessions following treatment

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of California, San Diego (UCSD) - Moores Cancer Center, La Jolla, California
  - University of Florida (UF) - Shands Cancer Center, Gainesville, Florida
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - University of Massachusetts, Worcester, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - John Theurer Cancer Center At Hackensack UMC, Hackensack, New Jersey
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University - Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sukhtankar DD, Fung JJ, Kim MN, Cayton T, Chiou V, Caculitan NG, Zalicki P, Kim S, Jo Y, Kim S, Lee JM, Choi J, Mun S, Chin A, Jang Y, Lee JY, Kim G, Kim EH, Huh WK, Jeong JY, Seen DS, Cardarelli PM. GPC-100, a novel CXCR4 antagonist, improves in vivo hematopoietic cell mobilization when combined with propranolol. PLoS One. 2023 Oct 25;18(10):e0287863. doi: 10.1371/journal.pone.0287863. eCollection 2023. PMID 37878624